CLINICAL TRIAL: NCT07201948
Title: Community Team Lifestyle Immersion Program for Chronic Disease Prevention and Control
Brief Title: Team Lifestyle Immersion Hypertension Control Project
Acronym: TLIP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Meharry Medical College (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 25-02-1555; 5P50MD017347-04 (NIH)
Record Dates: First submitted 2025-05-07; First posted 2025-10-01 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-03

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Physical Fitness; Dietary Approaches To Stop Hypertension

STUDY DESIGN:
Intervention Model Description: Two Study Arms:
  1. . Team Group
  2. . Individual Group All participants will receive the same intervention, but will be randomized into two study arms.
  Team Group: 4-6 participants will be assigned to work on their lifestyle as a team, motivating each other to adhere to the study intervention elements.
  Individual Group: Each participant will work on their own to adhere to the study intervention elements.
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Team Group (Active Comparator): 4-6 participants will be assigned to a Team. They will be instructed to work together and motivate each other to adhere to the intervention components, to attend intervention activities, and meet lifestyle modification goals.
  They will receive the intervention knowledge and skills training from:
  * Dietician
  * Physical Fitness Trainer
  * cardiologist They will also receive other support to enhance their lifestyle immersion from the research team.
  Interventions: Behavioral: Lifestyle Immersion Intervention that will address Nutrition, Physical Fitness, and BP Self-Monitoring3 Elements:
- Individual Group (Active Comparator): Individual participants will be instructed to self-motivate to adhere to the intervention components, to attend intervention activities, and meet lifestyle modification goals.
  They will receive the intervention knowledge and skills training from:
  * Dietician
  * Physical Fitness Trainer
  * cardiologist They will also receive other support to enhance their lifestyle immersion from the research team.
  Interventions: Behavioral: Lifestyle Immersion Intervention that will address Nutrition, Physical Fitness, and BP Self-Monitoring3 Elements:

INTERVENTIONS:
Behavioral: Lifestyle Immersion Intervention that will address Nutrition, Physical Fitness, and BP Self-Monitoring3 Elements: — 1. : Two distinct groups will be enrolled:
     * Those diagnosed with hypertension: BP >=140/90, within the last 2 years.
     * Those with BP >=130/80. Not yet diagnosed with hypertension.
  2. . Intervention: Comprehensive and integrated intervention components
     * Implemented by 3 certified experts (Dietician, Fitness Trainer, Cardiologist)
     * Modules: Education, Demonstration, Practical skill development sessions.
  3. . Intervention is based on American Hearts Association Life's Simple 7. The nutrition aspect will follow the DASH Diet plan.
  Other Names: Life's Simple 7; DASH Diet

SUMMARY:
This project is focuses on reducing the risk and progression of hypertension among a population that records high incidence of hypertension and other chronic ailments such as heart disease, diabetes, kidney failure, and obesity, with similar control measures. Several clinical trials over the last five decades have emphasized the importance of supportive lifestyle modification in the control of chronic disease that include a healthy diet, physical activity, quitting tobacco use, reducing alcohol use to the minimum, self-management of the disease, and adequate sleep. Study participants will receive motivation and skill development support in additional to specific nutrition, physical fitness, and self-management counselling from certified experts. This intervention incorporates elements of the American Heart Association prescription for health, Life's Simple 7 (LS7) lifestyle modification, the Dietary Approaches to preventing Hypertension (DASH) eating plan.

After receiving these interventions, participants will be contacted at 3-months, 6-months, and 12-months for follow-up. They will complete similar surveys to be compared to determine impact on their hypertension.

This intervention is complementary to usual pharmaceutical hypertension management.

DETAILED DESCRIPTION:
African Americans continue to bear disproportionate chronic disease morbidity and mortality, and tend to report lower benefits from clinical trials that include lifestyle modifications in addition to pharmaceutical management. This project uses hypertension as an index case for other chronic ailments such as heart disease, diabetes, kidney failure, and obesity, especially as their control measures are similar. Several clinical trials over the last five decades have emphasized the importance of supportive lifestyle modification in the control of chronic disease that include a healthy diet, physical activity, quitting tobacco use, reducing alcohol use to the minimum, self-management of the disease, and adequate sleep. Although socioeconomic factors can impact disease management outcomes, African Americans may require additional motivational support to first accept the notion of change of lifestyle and to adhere to the changes that may be a major shift in their eating and exercise habits. The need to positively impact chronic disease, particularly hypertension, morbidity and morbidity in the African American population deserves both pharmaceutical and non-pharmaceutical approaches. This intervention incorporates elements of the American Heart Association prescription for health, Life's Simple 7 (LS7) lifestyle modification, the Dietary Approaches to Stop Hypertension (DASH) eating plan, provides the knowledge and skills necessary for success, and introduces the motivation boost of participating in teams of 4-6 participants. The primary intervention outcome is adherence to the seven elements of LS7, measured by LS7 Scores at enrollment, and at 6- and 12-months follow-up. Secondary outcomes will include changes in SBP/DBP, BMI, Waist girth, and A1C. The study shall compare Team versus Individual study arms for participants recruited and managed in the health center and the home settings separately and combined. Intermediate outcomes will include, and not limited to biomarkers such as urine sodium, serum Plasminogen activator inhibitor-1 (PAI-1) for hypertension, Interleukin 6 (IL6), and C-reactive protein (CRP) for obesity.

The goal is to enroll 220 participants, half from health institutions (Nashville General Hospital & Mathew Walker Comprehensive Health Center) and the other half from the community (MDHA residence, Health Fairs, Churches etc.). Half of the participants will be people already diagnosed with hypertension (BP 140/90 or higher, or on hypertension medication) and half will be those at increased risk of developing hypertension with BP measurement 130/80 and above.

The study will be implemented in three phases:

Phase 1: Health Behavior Assessment. Phase 2: Intervention Development. Phase 3: Intervention Effectiveness Evaluation.

Intervention:

Participants will complete the study survey and a food frequency questionnaire and enrollment. they will also provide 5ml venous blood sample for biomarker assay. They will complete the same surveys at follow-up at 6- and 12-months to provide data for evaluation effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Reside in Davidson and surrounding counties of Tennessee.
* At least 30 years old.
* At increased risk for developing hypertension (already diagnosed or a strong family history).
* Be able to consent.
* Not planning to move from this study area in 12 months after enrollment.

Exclusion Criteria:

* Does not reside in Davidson and surrounding counties.
* Less than 30 years old, or older than 80 years.
* Not at assessed increased risk for hypertension.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2027-12-30 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Systolic and Diastolic Blood Pressure Change | 6 months & 12 months.
  Systolic and Diastolic blood pressure change will be computed as:
  SBP (enrollment) - SBP (Follow-up) DBP (enrollment) - DBP (Follow-up)

CONTACTS AND LOCATIONS:
Overall Officials: Flora Ukoli, MD, MPH, Study Director — Meharry Medical College; Stephena Miller-Hughes, Ph.D., Study Director — Meharry Medical College
Locations (1):
- Meharry Medical College, Nashville, Tennessee, United States